CLINICAL TRIAL: NCT04325594
Title: Optimization of the Complex Treatment of Nonischemic Dilated Cardiomyopathy Due to the Addition to the Standard Drug Therapy of Intracoronary Administration of Umbilical Cord-derived Mesenchymal Stromal Cells
Brief Title: The Application of the Umbilical Cord Mesenchymal Stem Cells in the Complex Treatment of Non-ischemic Heart Failure
Acronym: RegenHeart
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Research-Clinical Center for Cardiac Surgery and Transplantology LLP (Other)
Collaborators: State-Financed Health Facility "Samara Regional Medical Center Dinasty" (Other)
Responsible Party: Principal Investigator, Azkhojayev Aziz, MD, Cardiac surgeon, The Research-Clinical Center for Cardiac Surgery and Transplantology LLP
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCCCT 02-02-2020
Record Dates: First submitted 2020-03-03; First posted 2020-03-27 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chronic Heart Failure; Non-ischemic Cardiomyopathy; Non-ischemic Dilated Cardiomyopathy
Keywords: Chronic heart failure; Non-ischemic Cardiomyopathy; Non-ischemic Dilated Cardiomyopathy; Mesenchymal stromal cells; Umbilical cord; Regenerative Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Patients with chronic non-ischemic heart failure received a single intracoronary administration of 1×10⁷ umbilical cord-derived MSCs and continued optimal pharmacological therapy.
  Interventions: Biological: Intracoronary administration of umbilical cord-derived MSCs

INTERVENTIONS:
Biological: Intracoronary administration of umbilical cord-derived MSCs — A suspension of 1×10⁷ umbilical cord-derived mesenchymal stromal cells in 20 ml of heparinized saline was administered by intracoronary infusion into the left coronary artery via a standard 6 Fr catheter over 10 minutes (2 ml/min). The infusion was performed without balloon occlusion or interruption of coronary blood flow.

SUMMARY:
The purpose of this prospective single-arm clinical study was to evaluate the safety and potential efficacy of intracoronary administration of allogeneic umbilical cord-derived mesenchymal stromal cells (MSCs) as an addition to standard medical therapy in patients with chronic non-ischemic heart failure.

DETAILED DESCRIPTION:
This prospective, open-label, single-arm clinical trial investigated the safety and potential efficacy of intracoronary administration of allogeneic umbilical cord-derived mesenchymal stromal cells (MSCs) in patients with chronic non-ischemic heart failure.

A total of 30 patients were enrolled. All participants received standard pharmacological therapy and underwent a single intracoronary infusion of 1×10⁷ MSCs delivered into the left coronary artery during routine cardiac catheterization. The primary objective was to assess the safety of the cell therapy over the first 5 days of hospitalization. Secondary outcomes included changes in left ventricular ejection fraction (LVEF), end-diastolic and end-systolic volumes and diameters, serum NT-proBNP levels, NYHA functional class, 6-minute walk test distance, and quality of life indicators (SF-12, KCCQ, MLHFQ) at 1, 3, and 6 months post-infusion.

Although the study was originally registered with a control group and randomization, it was ultimately conducted as a single-arm design due to ethical and logistical constraints in recruitment. All patients received the same intervention, and no allocation or randomization was performed.

While most patients had clinical indications for an implantable cardioverter-defibrillator (ICD) in accordance with international guidelines, not all had the device implanted due to personal refusal of the procedure. Therefore, ICD presence was not required for inclusion in the study.

Although remuscularization of the myocardium was not a predefined endpoint, retrospective analysis revealed post-treatment thickening of the left ventricular posterior wall and interventricular septum in a subset of patients, as observed on cardiac computed tomography. This structural change was associated with improved systolic function and may guide future hypothesis-driven research.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and older
* Registered at the Research-Clinical Center for Cardiac Surgery and Transplantology
* Established diagnosis of non-ischemic dilated cardiomyopathy (NYHA Class III-IV)
* Non-ischemic etiology confirmed by coronary angiography or contrast-enhanced cardiac CT
* Left ventricular ejection fraction (LVEF) ≤ 35% based on echocardiography or cardiac CT
* Clinical indications for implantation of an implantable cardioverter-defibrillator (ICD), regardless of actual implantation status
* No clinical or laboratory signs of dysfunction or insufficiency of other major organs
* No history of malignancy within the past 5 years and no abnormal tumor markers
* Signed written informed consent

Exclusion Criteria:

* Ischemic heart disease or prior cardiac surgery, including coronary artery stenting
* Significant valvular heart disease, intracardiac thrombus, left ventricular aneurysm, hypertrophic, postpartum, alcoholic or restrictive cardiomyopathy, congenital heart defects, or resistant hypertension
* Stroke within the past 2 years
* Autoimmune or immunodeficiency disorders
* Polyvalent allergy
* Decompensated chronic comorbidities
* Use of systemic corticosteroids, cytotoxic or immunosuppressive drugs (e.g., cyclophosphamide, methotrexate, cyclosporine, azathioprine) within 4 weeks before enrollment
* Positive tests for hepatitis B or C, syphilis, or HIV/AIDS
* Active systemic infections requiring targeted antibiotic therapy
* Untreated peptic ulcer disease or history of gastrointestinal bleeding
* Clinically significant traumatic brain injury requiring treatment
* Uncontrolled epileptic seizures
* Porphyria
* Requirement for hospice-level care
* Alcohol or drug abuse, lack of permanent residence, severe depression, disorientation, or inability to participate in follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ischemic and arrhythmic events, abnormal laboratory and ECG findings within 5 days after intracoronary infusion of umbilical cord-derived MSCs [Safety Assessment] | First 5 days after infusion
  Safety will be assessed during a 5-day hospitalization period. Cardiac monitoring will be performed during and after intracoronary MSC infusion. Assessment includes incidence of ECG changes (e.g., ST-segment deviation), cardiac enzyme elevations (AST, ALT), local hypokinesia by echocardiography, and occurrence of ventricular arrhythmias. Laboratory evaluations include complete blood count, biochemistry, coagulation, and urinalysis on day 1 and day 5. Immune status will be assessed via neutrophil count and activity. Patients will be monitored in the intensive care unit for the first 24 hours.

SECONDARY OUTCOMES:
Change in left ventricular structure and function | 1, 3, and 6 months
  Changes in left ventricular ejection fraction (LVEF), end-diastolic and end-systolic volumes (EDV/ESV), and end-diastolic and end-systolic diameters (EDD/ESD), assessed by transthoracic echocardiography and cardiac computed tomography.
Change in NT-proBNP levels | 1, 3, and 6 months
  Serum levels of NT-proBNP as a biomarker of myocardial dysfunction.
Change in 6-minute walk test distance | 1, 3, and 6 months
  Functional capacity evaluated by the distance covered in the 6-minute walk test.
Change in NYHA functional class | 1, 3, and 6 months
  Heart failure severity graded by the New York Heart Association classification.
Change in quality of life | 1, 3, and 6 months
  Quality of life assessed using the SF-12 Health Survey, Kansas City Cardiomyopathy Questionnaire (KCCQ), and Minnesota Living with Heart Failure Questionnaire (MLHFQ).

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Azkhojayev, MD, Principal Investigator — The Research-Clinical Center for Cardiac Surgery and Transplantology LLP
Locations (1):
- The Research-Clinical Center for Cardiac Surgery and Transplantology LLP, Taraz, Zhambyl Oblysy, Kazakhstan

IPD SHARING:
Plan to Share IPD: No